CLINICAL TRIAL: NCT01124851
Title: A Multiple Dose Study of the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of ABT-652 Administered Once Daily to Subjects With an Excessive Daytime Sleepiness Disorder
Brief Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of ABT-652 in Subjects With Excessive Daytime Sleepiness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Hana Florian, MD/Associate Medical Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M11-685
Record Dates: First submitted 2010-04-26; First posted 2010-05-17 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Sleep Disorder
Keywords: Sleep disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): ABT-652 Dose 1 vs placebo capsules administered orally once daily for 7 days
  Interventions: Drug: ABT-652; Drug: Placebo
- Arm 2 (Experimental): ABT-652 Dose 2 vs placebo capsules administered orally once daily for 7 days
  Interventions: Drug: ABT-652; Drug: Placebo
- Arm 3 (Experimental): ABT-652 Dose 3 vs placebo capsules administered orally once daily for 7 days
  Interventions: Drug: ABT-652; Drug: Placebo

INTERVENTIONS:
Drug: ABT-652 — See arm description for details
Drug: Placebo — See arm description for details

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the drug ABT-652 given once daily to people with excessive daytime sleepiness. Subjects will be randomized to either ABT-652 or placebo in three sequential dosing groups for a 1-week treatment period.

ELIGIBILITY:
Inclusion Criteria

* Has current diagnosis of an excessive daytime sleepiness disorder, including narcolepsy, idiopathic hypersomnia, and obstructive sleep apnea
* Age 18 to 60 years Exclusion Criteria
* Has significant suicidal ideation
* Has a history of substance abuse
* Has a history of a certain significant medical conditions, including uncontrolled psychiatric diseases or disorders
* Use of certain medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Laboratory Tests | Baseline period to end of 1-week treatment period.
ECG | Baseline period to end of 1-week treatment period.
Adverse Events | Baseline period till 30 days after the last dose.
Vital Signs | Baseline period to end of 1-week treatment period.

SECONDARY OUTCOMES:
Maintenance Wakefulness Test | Baseline period to end of 1-week treatment period.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Site Reference ID/Investigator# 43241, Phoenix, Arizona
  - Site Reference ID/Investigator# 38092, Glendale, California
  - Site Reference ID/Investigator# 43264, San Diego, California
  - Site Reference ID/Investigator# 40402, New York, New York
  - Site Reference ID/Investigator# 38122, Durham, North Carolina